CLINICAL TRIAL: NCT04394117
Title: Controlled evaLuation of Angiotensin Receptor Blockers for COVID-19 respIraTorY Disease
Acronym: CLARITY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11052020
Record Dates: First submitted 2020-05-18; First posted 2020-05-19 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Coronavirus Disease 2019; COVID-19
Keywords: Angiotensin Receptor Blocker (ARB); Angiotensin Converting Enzyme 2 (ACE2); Coronavirus Disease 2019 (COVID-19); Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-Cov-2)
MeSH Terms: conditions — COVID-19 | interventions — Angiotensin Receptor Antagonists; candesartan; eprosartan; Irbesartan; Losartan; olmesartan; Telmisartan; Valsartan

STUDY DESIGN:
Intervention Model Description: CLARITY is a randomised control trial of two parallel groups;
  1. Standard Care + Angiotensin Receptor Blocker (ARB)
  2. Standard Care
  Participants will be randomised in a 1:1 ratio. Randomisation will be stratified according to country and whether the participant is planned for hospital admission or home-based care.
Who Masked: Outcomes Assessor
Masking Description: Trial Statistician and sponsor staff will remain blinded to treatment allocation throughout the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care + Angiotensin Receptor Blocker (ARB) (Active Comparator): Participants will receive an Angiotensin Receptor Blocker on top of the standard care provided by their institution.
  Interventions: Drug: Angiotensin Receptor Blockers
- Standard Care + Placebo (Placebo Comparator): Participants will receive a placebo on top of the standard care provided by their institution.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Angiotensin Receptor Blockers — Angiotensin Receptor Blockers (ARBs) have been in clinical use for more than 30 years for their cardiac and renal protective effects. ARBs mechanism of action is through selective inhibition of angiotensin-II (Ang-II) by competitive antagonism of the angiotensin receptor. ARBs displace ang-II from the angiotensin I receptor and produce their protective effects by reducing the downstream effects of ang-II induced vasoconstriction, aldosterone release, catecholamine release, arginine vasopressin release, water intake, and hypertrophic response The virus causing COVID-19, SARS-CoV-2, binds to the extracellular portion of Angiotensin-Converting-Enzyme-2 (ACE2) expressed on type II alveolar cells in the lungs which is followed by internalization of ACE2 before downregulating membrane ACE2 expression. Both these components appear to require angiotensin receptor Type 1 (AT1R), and ARBs, which block the actions of AT1R, would reduce the severity of COVID-19 and reduce the duration of symptoms
  Other Names: Candesartan; Eprosartan; Irbesartan; Losartan; Olmesartan; Telmisartan; Valsartan
  Arms: Standard Care + Angiotensin Receptor Blocker (ARB)
Other: Placebo — Placebo
  Arms: Standard Care + Placebo

SUMMARY:
The Controlled evaLuation of Angiotensin Receptor Blockers for COVID-19 respIraTorY disease (CLARITY) study is a pragmatic prospective, open-label, randomised controlled trial. CLARITY aims to examine the effectiveness of angiotensin II receptor blockers (ARBs) on improving the outcomes of people who tested positive for COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

Potential participants must satisfy all of the following:

1. Laboratory-confirmed* diagnosis of Severe Acute Respiratory Syndrome-Coronavirus-2 infection within 10 days prior to randomisation
2. Age ≥ 18 years
3. a) Systolic Blood Pressure (SBP) ≥ 120 mmHg OR b) SBP ≥ 115 mmHg and currently treated with a non-Renin Angiotensin Aldosterone System inhibitor Blood Pressure (BP) lowering agent that can be ceased
4. Participant and treating clinician are willing and able to perform trial procedures.
5. Either Intended for hospital admission for management of COVID-19, or (In Australia Only) Intended for management at home with one or more of the following criteria:

   1. Age≥60 years
   2. Body Mass Index ≥30kg/m2 (derived from the patient's self-report of their height and weight where these are not measured directly)
   3. Diagnosis of diabetes defined as HbA1c ≥7% and/or the consumption of glucose lowering medication
   4. History of cardiovascular disease
   5. History of chronic respiratory illness
   6. Currently treated with immunosuppression

Exclusion Criteria:

1. Currently treated with an angiotensin-converting enzyme inhibitor, Angiotensin Receptor Blocker or aldosterone antagonist, aliskiren, or angiotensin receptor-neprilysin inhibitors (ARNi)
2. Serum potassium > 5.2 mmol/L or no potassium testing within the last 3 months
3. For those intended for hospital admission, an estimated Glomerular Filtration Rate (eGFR) <30ml/min/1.73m2 or no eGFR testing within the last 3 months, or For those intended for management at home (Australia only), an eGFR <45ml/min/1.73m2 or no eGFR testing within the last 3 months
4. Known symptomatic postural hypotension
5. Known biliary obstruction, known severe hepatic impairment (Child-Pugh-Turcotte score 10-15) - see Table below
6. Intolerance of ARB
7. Pregnancy or risk of pregnancy, defined as;

   1. (In Australia only) Women younger than 51 years who have not had a negative pregnancy test during the past 3 days and/or who do not agree to use adequate contraception
   2. (In India Only) Women who are pregnant
8. Women who are currently breastfeeding
9. Individuals who are not able to take medications by mouth at enrolment, or who are not expected to be able to take medications by mouth during the first 48 hours after randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
7-Point National Institute of Health Clinical Health Score | 14 Days
  To determine whether the addition of the intervention, compared to standard care, changes the clinical health score of a participant on the following scale;
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO);
  7. Death;

SECONDARY OUTCOMES:
7-Point National Institute of Health Clinical Health Score | 28 Days
  To determine whether the addition of the intervention, compared to standard care, changes the clinical health score of a participant on the following scale;
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO);
  7. Death;
Mortality | 28 Days
  To determine whether the addition of the intervention, compared to standard care, changes the risk of all cause mortality
Mortality | 90 Days
  To determine whether the addition of the intervention, compared to standard care, changes the risk of all cause mortality
Intensive Care Unit Admission | 28 Days
  To determine whether the addition of the intervention, compared to standard care, changes the count of all cause Intensive Care Unit admission
Intensive Care Unit Admission | 90 Days
  To determine whether the addition of the intervention, compared to standard care, changes the count of all cause Intensive Care Unit admission
Intensive Care Unit Number of Days | 90 Days
  To determine whether the addition of the intervention, compared to standard care, changes the number of days total, of intensive care unit admission
Respiratory Failure | 28 Days
  To determine whether the addition of the intervention, compared to standard care, changes the incidence of respiratory failure
Dialysis Requirement | 28 Days
  To determine whether the addition of the intervention, compared to standard care, changes the requirements for dialysis
Hospitalisation Days | 28 Days
  To determine whether the addition of the intervention, compared to standard care, changes the number of hospitalisation days
Hospitalisation Days | 90 Days
  To determine whether the addition of the intervention, compared to standard care, changes the number of hospitalisation days
Ventilator-Free Days | 28 Days
  To determine whether the addition of the intervention, compared to standard care, changes need for ventilation
Dialysis Days | 28 Days
  To determine whether the addition of the intervention, compared to standard care, changes need for dialysis
Acute Kidney Injury | 28 Days
  To determine whether the addition of the intervention, compared to standard care, changes risk of acute kidney injury, based on the Kidney Disease: Improving Global Outcomes definition
Hypotension Requiring Vasopressors | 28 Days
  To determine whether the addition of the intervention, compared to standard care, changes risk of hypotension requiring vasopressors

OTHER OUTCOMES:
Hyperkalaemia | Day 28
  To determine whether the addition of the intervention, compared to standard care, changes risk of hyperkalaemia.
Oxygen Saturation | Day 28
  To determine whether the addition of the intervention, compared to standard care, changes risk of decreased oxygen saturation
Oxygen Saturation | Day 14
  To determine whether the addition of the intervention, compared to standard care, changes risk of decreased oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Meg Jardine, Study Chair — University of Sydney
Locations (22):
- Australia (15):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Canterbury Hospital, Campsie, New South Wales
  - The Sutherland Hospital, Caringbah, New South Wales
  - Concord Hospital, Concord, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Northern Health, Epping, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria
  - Western Health, St Albans, Victoria
- India (7):
  - Government Medical College & Hospital, Chandigarh
  - Post Graduate Institute of Medical Education & Research, Chandigarh
  - Lok Nayak Jai Prakash, Delhi
  - Kasturba Medical College, Manipal
  - Christian Hospital, Nowrangapur
  - Jivenrekha Hospital, Pune
  - All India Institute of Medical Science, Raipur

IPD SHARING:
Plan to Share IPD: Yes
Trial data will be disseminated in the form of a publication to a relevant clinical journal and presentation at appropriate scientific conferences.
  Individual participant data that underlie the results reported, after de-identification (text, tables, figures, and appendices), may be shared with Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: To be confirmed
Access Criteria: To be determined

REFERENCES:
- [Derived] Jardine MJ, Kotwal SS, Bassi A, Hockham C, Jones M, Wilcox A, Pollock C, Burrell LM, McGree J, Rathore V, Jenkins CR, Gupta L, Ritchie A, Bangi A, D'Cruz S, McLachlan AJ, Finfer S, Cummins MM, Snelling T, Jha V; CLARITY trial investigators. Angiotensin receptor blockers for the treatment of covid-19: pragmatic, adaptive, multicentre, phase 3, randomised controlled trial. BMJ. 2022 Nov 16;379:e072175. doi: 10.1136/bmj-2022-072175. PMID 36384746
- [Derived] McGree JM, Hockham C, Kotwal S, Wilcox A, Bassi A, Pollock C, Burrell LM, Snelling T, Jha V, Jardine M, Jones M; CLARITY Trial Steering Committee. Controlled evaLuation of Angiotensin Receptor Blockers for COVID-19 respIraTorY disease (CLARITY): statistical analysis plan for a randomised controlled Bayesian adaptive sample size trial. Trials. 2022 Apr 27;23(1):361. doi: 10.1186/s13063-022-06167-2. PMID 35477480
- [Derived] Hockham C, Kotwal S, Wilcox A, Bassi A, McGree J, Pollock C, Burrell LM, Bathla N, Kunigari M, Rathore V, John M, Lin E, Jenkins C, Ritchie A, McLachlan A, Snelling T, Jones M, Jha V, Jardine M; CLARITY Investigators. Protocol for the Controlled evaLuation of Angiotensin Receptor blockers for COVID-19 respIraTorY disease (CLARITY): a randomised controlled trial. Trials. 2021 Aug 28;22(1):573. doi: 10.1186/s13063-021-05521-0. PMID 34454580